CLINICAL TRIAL: NCT00202579
Title: Evaluation of the Effects on Peripheral and Central Haemodynamics Parameters, Safety, and Tolerance of Three-hour Intravenous Perfusion (0.1 mg/kg) of Ivabradine Given to Severe Congestive Heart Failure Patients
Brief Title: Efficacy and Safety of Ivabradine in Severe Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CL2-16257-053
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

INTERVENTIONS:
Drug: Ivabradine

SUMMARY:
To evaluate the effects on heart function of ivabradine administered to patients with severe chronic heart failure

ELIGIBILITY:
Inclusion Criteria:

* systolic congestive heart failure
* sinus rhythm, HR >= 80bpm

Exclusion Criteria:

* unstable cardiovascular condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-09; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Haemodynamic parameters
Twelve-lead ECG
Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Echocardiography
Neurohormones

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tavazzi, Pr, Study Chair — Policlinico San Matteo
Locations (1):
- Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com